CLINICAL TRIAL: NCT00716664
Title: Pilot Study: Do Physiotherapy Musculoskeletal Techniques Improve Forced Expiratory Volume in One Second in Adults With Cystic Fibrosis?
Brief Title: Do Musculoskeletal Techniques Improve Forced Expiratory Volume in One Second in Adults With Cystic Fibrosis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Mrs Catherine Sandsund, Honorary Research Fellow in Physiotherapy,, Department of Cystic Fibrosis, Royal Brompton Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06/Q0404/81
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2008-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; musculoskeletal; exercise capacity; posture; lung function; physical functioning
MeSH Terms: conditions — Cystic Fibrosis | interventions — Musculoskeletal Manipulations; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): The experimental group receives the intervention in addition to normal optimal care
  Interventions: Other: A treatment series of gentle joint and muscle movements
- 2 (Active Comparator): The active comparator, or control group, receives normal optimal care only
  Interventions: Other: Control group measurements

INTERVENTIONS:
Other: A treatment series of gentle joint and muscle movements — Undertaken by a physiotherapist, weekly, for six weeks
  Other Names: manual therapy; physical therapy; mobilisation; musculoskeletal techniques
  Arms: 1
Other: Control group measurements — The control group are measured using the same outcome measures at the same time intervals, but receive no active intervention
  Arms: 2

SUMMARY:
The pilot study aims to evaluate the effects of a treatment series of gentle joint and muscle movements (in addition to normal optimal care)on lung function, exercise capacity and posture in stable adults with cystic fibrosis.

DETAILED DESCRIPTION:
Study type:

Prospective, single-blinded, randomised control trial

Consent

* Prospective subjects will be given written and verbal information about the project and will be given at least 24 hours to consider entry to the study.
* Subjects will give written consent to participate in the project. The top copy will be included in the patient's medical record and a copy placed in the patient's study file.
* A letter will be written to the subject's General Practitioner outlining the purpose of the study and inviting him/her to make contact to discuss the study in more detail if there are any queries or concerns.
* At the time of consent, the appointments for the duration of the interventions and potential follow-up will be made.

Intervention for the treatment group A treatment series of gentle joint and muscle movements (musculoskeletal interventions) will be undertaken by a physiotherapist, weekly, for six weeks. A chaperone would be available if requested by the subject (the patients would be made aware of this when informed about the study.)

Proposed Interventions

The physiotherapy musculoskeletal assessment and intervention may last up to one hour and may include one or a combination of the following techniques which are well described in populations with postural changes, thoracic stiffness, discomfort and/or pain:

* Specific, gentle oscillatory mobilisations to the rib cage and thoracic spine of the subjects to improve joint alignment and mobility, and to reduce pain. These techniques should optimise chest wall mechanics, improving the length-tension relationships of the muscles and normalising movement to dysfunctional areas (Maitland et al. 2001; Mulligan 2005).
* Treatment of specific muscle dysfunction or tight muscle groups to further optimise muscle length and biomechanical relationships in the area (Massery 2005), leading to improved efficiency of recruitment and improved power output (Travell & Simons 1983).
* Neural stretches consisting of specific stretches to the neural system, to improve the neural dynamics aiming to reduce symptoms, increase range of motion and optimise nerve conduction in order to normalise the working relationship of the joint and muscular components of the area (Butler 1991).
* Neuromuscular techniques restore normal movement through facilitation. Guidance by the hands of the physiotherapist inhibits abnormal activity and facilitates a more optimal muscular activity. Specific postural awareness exercises are used to educate and re-establish normal movement, augmenting gains made with treatment (Carr & Shepherd 1998).
* Home programme to reinforce the progress during the treatment sessions consisting of no more than three specific stretching or strengthening exercises.

Control Group The control group would be invited to undertake the measurements at similar time intervals to the treatment group (0, 3, 6 and 12 weeks). They will receive their usual care but no placebo intervention. The control group would be offered treatment after the completion of data collection for the study, if the intervention is shown to be beneficial.

Potential Benefits

* Improvement in lung function
* Improved thoracic excursion
* Reduction in chest wall pain
* Improvement in exercise capacity. Potential risks
* Post treatment soreness lasting up to 24 hours.
* In the event of undetected exclusion criteria there is the potential for a rib fracture.
* There may be a relative or transient risk of syncopal event or vagal stimulation.

Data Collection The outcome measures will be undertaken by an independent observer to pre-agreed protocols, before the first intervention session (Week 0) and after the third (Week 3) and sixth treatments (Week 6). Full lung function will be repeated at the end of the intervention period. The outcome measurements will be repeated at six weeks (Week 12) following the end of treatment to explore the sustainability of any treatment effects. On completion of or withdrawal from the study, subjects will be invited to complete an exit interview questionnaire.

Proposed Primary Outcome measure

* Forced expiratory volume in one second (FEV1). Secondary Outcome Measures
* Forced vital capacity (FVC), peak expiratory flow rate (PEFR)
* Visual analogue scale for pain (Huskisson 1974)
* Modified shuttle test (Bradley et al. 1999) monitoring oxygen saturation and heart rate and Borg CR10 scale of perceived exertion (Borg 1982).
* The Cystic Fibrosis Quality of Life Questionnaire, section one: physical functioning - Questionnaire I (Gee et al. 2000)
* Flexi curve measurements of posture (Tillotson & Burton 1991)
* Chest wall excursion measurements (LaPier & Cook 2000)
* Full lung function will be measured ≤ one month prior to the start of the study and at the end of the intervention period
* Questionnaire II - the subject's perspective.

Statistical Analysis and reporting The statistical analysis has been discussed with Mr Michael Roughton, Statistician, Royal Brompton Hospital and Imperial College London.

Sample size calculation As there is no recent similar study available upon which to base a sample size calculation this will be a pilot study. The study aims to recruit 10 to the treatment group and 10 to the control group.

Statistical analysis The quantitative outcomes will be analysed using the Mann-Whitney test (assuming that this small set of data will not be normally distributed) to test for any difference for each variable from baseline; and will be analysed at each assessment point to establish the most beneficial length of treatment and the sustainability of any effects. The results will be represented graphically and in tables.

In the event of any missing data, withdrawal or non-compliance the patients will be analysed as 'intention to treat'.

Subjects will be allocated using "the method of minimisation" (Evans, Day, & Royston) to either the control or treatment group. This method weights a number of prognostic factors and their potential influence upon the outcome (e.g. FEV1 severity, sex of the subject). Two prognostic factors will be used reducing the predictability of which group hey will be allocated to.

The subjects are then allocated using the method of minimisation using a computer generated randomisation schedule running a minimisation algorithm thus ensuring a greater chance of a subject being allocated to a group that will optimise the comparability of the groups since the number of subjects being studied is small, but with the allocation still being subject to randomisation principles. The randomisation will be carried out by an independent member of the Department of Cystic Fibrosis and concealed from the independent observer.

Adverse events Any adverse events will be documented in the patient's medical notes, discussed with the medical staff and reported to the Chairman of the Ethics Committee.

Data Protection Patient data will be coded to protect their identities. Written data will be kept in a locked filing area within the Department of Cystic Fibrosis, Royal Brompton Hospital. Data analysis will be done on a password protected computer. Back-up will be maintained on a CD-ROM in a locked filing area within the Department of Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Reported postural changes, stiffness, discomfort and/or pain of musculoskeletal origin in the thoracic spine or chest wall.
* Diagnosis of cystic fibrosis (confirmed by genotype or a sweat sodium concentration of >70mmol/l or sweat chloride of >60mmol/l)
* Sixteen years of age or over
* Patients in a stable clinical state with lung function at the time of entry that is within 10% of the mean of the last two recordings (separated by at least one month).
* Forced Expiratory Volume in 1 second (FEV1) ≥30% predicted at time of entry to the study.

Exclusion Criteria:

* Evidence of a current respiratory exacerbation (worsening) as defined by Thornton et al. 2004
* Cor pulmonale (right heart failure)
* Low bone density (Z score < -3)(WHO Study Group 1994)
* Previous history of spontaneous fractures
* Past history of spinal fracture or other known arthropathic (joint) or spinal disease process
* Currently undergoing musculoskeletal (physiotherapy, chiropractic or osteopathic) treatment
* Pregnancy
* Inability to give consent
* Current enrollment in another research trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second | 12 weeks

SECONDARY OUTCOMES:
Forced vital capacity, peak expiratory flow rate | 12 weeks
Visual analogue scale for pain | 12 weeks
Modified shuttle test | 12 weeks
The Cystic Fibrosis Quality of Life Questionnaire, section one: physical functioning | 12 weeks
Flexi curve measurements of posture | 12 weeks
Chest wall excursion measurements | 12 weeks
Full lung function will be measured ≤ one month prior to the start of the study and at the end of the intervention period | 12 weeks
Questionnaire II - the subject's perspective | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton Hospital, London, London, United Kingdom